CLINICAL TRIAL: NCT07322926
Title: Is It So Hard To Predict Complicated Diverticulitis?
Status: Completed | Type: Observational
Sponsor: Haydarpasa Numune Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Naz Tayyar, Resident, Haydarpasa Numune Training and Research Hospital
Other Study IDs: HaydarpasaNumune
Record Dates: First submitted 2025-11-24; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-11

CONDITIONS: Diverticulitis
Keywords: Diverticulitis; neutrophil-to-lymphocyte ratio; lymphocyte-to-monocyte ratio; emergency
MeSH Terms: conditions — Diverticulitis; Emergencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with left colonic diverticulitis: no intervention

SUMMARY:
Is It So Hard To Predict Complicated Diverticulitis?

Objective: Acute diverticulitis (AD) is a frequent cause of abdominal pain leading to emergency department visits. Many biomarkers have been identified to predict the risk of developing complicated diverticulitis. In our study, we aimed to reveal the sensitivity of these biomarkers in order to better differentiate uncomplicated AD from complicated ones.

Methods: 101 patients who were diagnosed with AD in the emergency outpatient clinic between 2018 and 2022, registered in the database of our hospital, were evaluated retrospectively. Demographic data of the patients and laboratory results at the time of admission were evaluated. Patients were classified as having non-complicated (Group I) or complicated diverticulitis (Group II) based on the World Society of Emergency Surgery (WSES) criteria. Laboratory values at admission, including albumin, white blood cell count (WBC), C-reactive protein (CRP), neutrophil count, neutrophil-to-lymphocyte ratio (NLR), and lymphocyte-to-monocyte ratio (LMR), were evaluated.

DETAILED DESCRIPTION:
101 patients who were diagnosed with AD in the emergency outpatient clinic between 2018 and 2022, registered in the database of our hospital, were evaluated retrospectively. Demographic data of the patients and laboratory results at the time of admission were evaluated. Patients were classified as having non-complicated (Group I) or complicated diverticulitis (Group II) based on the World Society of Emergency Surgery (WSES) criteria. Laboratory values at admission, including albumin, white blood cell count (WBC), C-reactive protein (CRP), neutrophil count, neutrophil-to-lymphocyte ratio (NLR), and lymphocyte-to-monocyte ratio (LMR), were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the Haydarpaşa Numune Training and Research Hospital General Surgery Clinic
* First episode of acute diverticulitis
* Diagnosis confirmed by contrast-enhanced abdominal computed tomography (CT)
* Admission between 2018 and 2022
* Retrospective identification from the hospital registry system

Exclusion Criteria:

* Recurrent episodes of diverticulitis
* History of prior colorectal surgery
* Symptom duration longer than 7 days before admission
* Inconsistent physical examination findings with laboratory or imaging results
* Age under 18 years
* Pathologically confirmed malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 101 patients who were admitted to the Haydarpaşa Numune Training and Research Hospital General Surgery Clinic with the diagnosis of first acute diverticulitis attack between the years 2018-2022 were chosen.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Number of participants diagnosed with complicated acute diverticulitis according to the WSES classification | Time frame is the length of stay usually between 1-14 days
  Acute diverticulitis severity will be classified using the World Society of Emergency Surgery (WSES) diverticulitis grading system based on contrast-enhanced abdominal computed tomography (CT) findings at the time of admission.
  Patients will be categorized as having uncomplicated diverticulitis (WSES grades 1a and 1b) or complicated diverticulitis (WSES grades 2, 3, and 4). The primary outcome is the number of participants diagnosed with complicated diverticulitis.

CONTACTS AND LOCATIONS:
Locations (1):
- Haydarpasa Numune Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chabok A, Andreasson K, Nikberg M. Low risk of complications in patients with first-time acute uncomplicated diverticulitis. Int J Colorectal Dis. 2017 Dec;32(12):1699-1702. doi: 10.1007/s00384-017-2912-7. Epub 2017 Oct 16. PMID 29038965
- [Result] Feingold D, Steele SR, Lee S, Kaiser A, Boushey R, Buie WD, Rafferty JF. Practice parameters for the treatment of sigmoid diverticulitis. Dis Colon Rectum. 2014 Mar;57(3):284-94. doi: 10.1097/DCR.0000000000000075. No abstract available. PMID 24509449
- [Result] Zaborowski AM, Winter DC. Evidence-based treatment strategies for acute diverticulitis. Int J Colorectal Dis. 2021 Mar;36(3):467-475. doi: 10.1007/s00384-020-03788-4. Epub 2020 Nov 6. PMID 33156365
- [Result] Biondo S, Golda T, Kreisler E, Espin E, Vallribera F, Oteiza F, Codina-Cazador A, Pujadas M, Flor B. Outpatient versus hospitalization management for uncomplicated diverticulitis: a prospective, multicenter randomized clinical trial (DIVER Trial). Ann Surg. 2014 Jan;259(1):38-44. doi: 10.1097/SLA.0b013e3182965a11. PMID 23732265